CLINICAL TRIAL: NCT06232304
Title: Transforming Behavioral Healthcare to Improve the Quality of Life for Individuals With Childhood-onset Lupus
Brief Title: Transforming Care for Individuals With Childhood-onset Systemic Lupus Erythematosus
Acronym: cSLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Hospital for Sick Children (Other); Seattle Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Tulane University (Other); University of Alabama at Birmingham (Other); Helen DeVos Children's Hospital (Other); Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Natoshia Cunningham, Associate Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009194
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus of Childhood (Disorder)
Keywords: lupus; depression; depressive symptoms; fatigue; pain; SLE; rheumatic disease; rheumatology; cognitive behavioral; Childhood-onset Systemic Lupus Erythematosus; cSLE; Implementation; Coping skills; Mindfulness
MeSH Terms: conditions — Depression; Fatigue; Pain; Rheumatic Diseases | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomization occurs at the site level. Participants enrolled will either receive TEACH, a coping skills program, or medical treatment as usual.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked to who received TEACH and who did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEACH (Experimental): Participants will undergo a cognitive behavioral coping skills program and continue medical treatment as usual.
  Interventions: Behavioral: TEACH
- Control (No Intervention): Participants will only continue medical treatment as usual.

INTERVENTIONS:
Behavioral: TEACH — TEACH is a cognitive behavioral coping skills program. It consists of six one-hour weekly sessions that are conducted either in-person or remotely.
  Other Names: Treatment and Education Approach for Childhood-onset Lupus
  Arms: TEACH

SUMMARY:
This study aims to investigate the feasibility and effectiveness of a cognitive behavioral coping skills program, Treatment and Education Approach for Childhood-onset Lupus (TEACH), for youth with cSLE when integrated into medical care. This TEACH program aims to teach participants skills in order to cope with fatigue, pain, and depressive symptoms--symptoms that commonly affect adolescents and young adults with lupus.

DETAILED DESCRIPTION:
Background/Rationale: Childhood-onset systemic lupus erythematosus (cSLE) is a chronic, multisystem, autoimmune disease that disproportionately impacts females of color. It is associated with a more severe disease presentation, and a 20-fold increased risk of mortality compared to adult-onset SLE. Depressive symptoms, anxiety, fatigue, and pain are among the most common presenting complaints which impact health-related quality of life (QOL) in individuals with cSLE. These symptoms are potentially modifiable with behavioral intervention. Our team has created an evidence-based, brief and tailored 6-session program, Treatment and Education Approach for Childhood-onset lupus [TEACH], which can be delivered in person or remotely using cognitive behavioral therapy (CBT) strategies to address mental health symptoms, fatigue, and pain. Our nearly completed multi-site RCT, comparing TEACH (delivered by research interventionists) to standard medical care, shows efficacy for psychological/functional outcomes and benefit for disease-related outcomes. Although TEACH is extremely promising, patients do not currently have access to this program as part of their rheumatology care. cSLE patients would likely benefit from TEACH integrated into their medical care, leveraging existing relationships with their providers. As rheumatology teams are often identified as primary providers by cSLE patients, they have a key role in facilitating mental health intervention to enhance patient QOL. They are therefore well-positioned for training in the management of these common, debilitating, yet modifiable symptoms.

Objective: The objective is to determine the effectiveness of a coping skills program, TEACH, designed to improve psychological/functional- and disease- related outcomes in youth with cSLE. We will also investigate longitudinal trajectories of depressive symptoms in recipients and explore implementation outcomes.

Specific Aims & Hypotheses:

Aim 1: To examine the effect of TEACH on psychological/ functional outcomes and disease-related outcomes in youth with cSLE in real-world rheumatology settings versus medical TAU at post assessment (after 8 weeks). We hypothesize that both psychological/functional outcomes (depressive symptoms [primary], fatigue [secondary], anxiety, pain, cognitive function) and disease-related outcomes (health-related QOL, medication adherence, disease activity/flares) will significantly improve for the TEACH group vs medical TAU.

Aim 2: To determine longitudinal trajectories (over 1 year) of depressive symptoms, the impact of TEACH, and its association with patient characteristics, psychological/functional outcomes, and disease-related outcomes. We hypothesize that: i) distinct trajectories of depressive symptoms [low stable, improving, worsening] will emerge through growth mixture modeling, ii) TEACH vs TAU will be associated with decreased depressive symptoms and improved functioning over time, and iii) worsening depressive symptoms will be associated with poorer psychological/functional outcomes & disease-related outcomes.

Aim 3: To evaluate TEACH implementation outcomes using a mixed method approach. We will identify implementation outcomes (e.g., barriers and facilitators, acceptability, fidelity, reach, sustainability) of TEACH through surveys and interviews of providers and patients to inform future adoption/sustainability. We hypothesize results will demonstrate TEACH implementation success (e.g., high acceptability, appropriateness, feasibility, fidelity, knowledge of intervention), and metrics of sustainability will be positive.

Research Strategy: We propose a multi-site stepped wedge trial utilizing an effectiveness-implementation hybrid design (type 1) to study the clinical effectiveness and implementation of TEACH administered by integrated trained mental health champions. Seven participating sites across the US and Canada will train integrated mental health champions on the rheumatology team to deliver an empirically supported coping skills program, TEACH, to youth with cSLE. Our multidisciplinary research team consists of rheumatologists, behavioral scientists, and consumer advocates representing several national lupus organizations. Impact: Integrated mental health champions will provide evidence-based strategies to improve psychologicaland disease-related outcomes in youth with cSLE. Our vision is to transform care and improve patient QOL.

ELIGIBILITY:
Inclusion Criteria:

* 1) be diagnosed with cSLE, meeting the revised American College of Rheumatology Classification Criteria for SLE by age 18 years
* 2) be between the ages of 12 and 22 years
* 3) in recognition of the heterogeneity of cSLE symptoms, have elevations in fatigue (i.e., T scores ≥60; or at least moderate symptoms, on the PROMIS measure) OR depressive symptoms (≥5 on the PHQ-9, T Score ≥ 60 on the BDI or CDI II ), OR pain (i.e., average pain ≥3 out of 10 on the Pain VAS)
* 4) have English language proficiency (their primary caregiver can have English or Spanish language proficiency for the child to enroll)
* 5) those under age 18 years (US), or 16 years (Canada) must have a consenting caregiver

Exclusion Criteria:

* 1) other chronic medical conditions (e.g., juvenile arthritis)
* 2) a documented developmental delay, severe cognitive impairment, or thought disorder
* 3) an untreated major psychiatric illness (e.g., bipolar disorder, psychosis, severe depression (PHQ9 score ≥21, BDI/CDI II > 90) or active suicidal ideation (SI), based on the Pediatric Health Questionnaire (PHQ-9) items plus clinical interview; see Measures section)

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms, as measured by the Children's Depression Inventory-2 (CDI-2) and Beck Depression Inventory-II (BDI-II) (primary) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The CDI-2 measures depressive symptoms on a scale of 0-54, with 0 indicating low levels of depressive symptoms, and 54 indicating high levels of depressive symptoms. The BDI-II measures depressive symptoms on a scale of 0 to 63, with 0 indicating low levels of depressive symptoms and 63 indicating high levels of depressive symptoms.
Depressive symptoms, as measured by the Patient Health Questionnaire - 9 (PHQ-9) (primary) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PHQ-9 measures depressive symptoms on a scale of 1-27, with 1 indicating low levels of depressive symptoms, and 27 indicating high levels of depressive symptoms.
Fatigue, as measured by the PROMIS Fatigue short form (secondary) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The adult PROMIS Fatigue SF measures fatigue one a scale of 10-40; 10 indicating no fatigue, 40 indicating high levels of fatigue. The pediatric PROMIS Fatigue SF measures on a scale of 0-40; 0 indicating no fatigue and 40 indicating high levels of fatigue.
Pain, as measured by the Pain Visual Analog Scale (VAS) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The Pain VAS measures three items on a scale of 0-10, with 0 indicating no pain and 10 indicating the worst possible pain.
Pain, as measured by PROMIS Pain Interference Short Form | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Interference due to pain symptoms over the past week will be collected from youth (0-32, where 0 indicates low levels of pain interference and 32 is the maximum score for pain interference) and adults (8-40, where 8 indicates low levels of pain interference and 40 is the maximum score for pain interference).
Psychological stress, as measured by the PROMIS psychological stress experience measure | T1 (baseline), T2 (8 weeks)
  PROMIS psychological stress experience measure is validated for pediatrics and adults. Scores range from 0-95 where 0 indicates no psychological stress and 95 is the maximum score for psychological stress.
Cognitive functioning, as measured by the PROMIS Cognitive Function Short Form for Adults and the PROMIS Cognitive Function Short Form for Pediatrics | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  PROMIS Cognitive Function Adult form scores range from 8-40, where 8 indicates never having cognitive dysfunction, and 40 indicates very often having cognitive dysfunction. PROMIS Cognitive Function Pediatric form scores range from 7-35, where 7 indicates never having cognitive dysfunction, and 35 indicates having cognitive dysfunction all of the time.
Quality of life, as measured by the Pediatric Quality of Life (PedsQL) Generic Core | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PedsQL measures quality of life in several aspects such as health, school, daily activities. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life.
Quality of life, as measured by the Pediatric Quality of Life (PedsQL) Rheumatology Core | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PedsQL measures quality of life in several aspects such as pain and hurt, daily activities, treatment, worry, and communication. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life.
Medication adherence, as measured by the Medication Adherence Self-Report Inventory (MASRI) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The MASRI measures medication adherence on a scale of 0%-100%, such that lower scores indicate less adherence and higher scores indicate more adherence.
Disease activity, as measured by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The SLEDAI 2K measures disease activity in SLE, and takes into consideration descriptors of the disease such as arthritis and vasculitis. Higher scores indicate more active disease/flares, and lower scores indicated less disease activity.
Disease activity, as measured by the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The SLICC measures disease activity by assessing descriptors in SLE. Higher scores indicate greater disease activity, lower scores indicate lesser disease activity
Disease activity, as measured by the Lupus Low Disease Activity State (LLDAS) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The LLDAS is a score from 0-5, where 0 indicates higher disease activity state and 5 indicates lower disease activity state. The LLDAS includes 5 components, each receiving either a 1 (true) or a 0 (false): 1. SLEDAI score less than or equal to 4, 2. no new lupus disease activity, 3. a SELENA-SLEDAI less than or equal to 1, 4. a maintained low prednisolone dose, and 5. well tolerated maintenance doses or immunosuppressive drugs and approved biological agents.
Disease manifestations | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Disease manifestation will be assessed by use of the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) criteria checklist.
Anxiety, as measured by the Screen for Child Anxiety Related Disorders (SCARED) and Screen for Adult Anxiety Related Disorders (SCAARED) | T1 (baseline), T2 (8 weeks)
  The SCARED measures anxiety in children on a scale of 0 to 82, such that lower scores indicates low levels of anxiety, and high scores indicated high levels of anxiety. The SCAARED measures anxiety in adults on a scale of 0 to 88 such that lower scores indicated lower levels of anxiety and high scores indicate higher levels of anxiety. Both scales are comprised of sub-scales to measure types of anxiety (such as separation anxiety).

SECONDARY OUTCOMES:
Depressive symptoms, as measured by the Children's Depression Inventory-2 (CDI-2) and Beck Depression Inventory-II (BDI-II) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The CDI-2 measures depressive symptoms on a scale of 0-54, with 0 indicating low levels of depressive symptoms, and 54 indicating high levels of depressive symptoms. The BDI-II measures depressive symptoms on a scale of 0 to 63, with 0 indicating low levels of depressive symptoms and 63 indicating high levels of depressive symptoms.
Depressive symptoms, as measured by the Patient Health Questionnaire - 9 (PHQ-9) (primary) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PHQ-9 measures depressive symptoms on a scale of 1-27, with 1 indicating low levels of depressive symptoms, and 27 indicating high levels of depressive symptoms.
Fatigue, as measured by the PROMIS Fatigue SF | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The adult PROMIS Fatigue SF measures fatigue one a scale of 10-40; 10 indicating no fatigue, 40 indicating high levels of fatigue. The pediatric PROMIS Fatigue SF measures on a scale of 0-40; 0 indicating no fatigue and 40 indicating high levels of fatigue.
Pain, as measured by the Pain Visual Analog Scale (VAS) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The Pain VAS measures three items on a scale of 0-10, with 0 indicating no pain and 10 indicating the worst possible pain.
Pain, as measured by PROMIS Pain Interference Short Form | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Interference due to pain symptoms over the past week will be collected from youth (0-32, where 0 indicates low levels of pain interference and 32 is the maximum score for pain interference) and adults (8-40, where 8 indicates low levels of pain interference and 40 is the maximum score for pain interference).
Psychological stress, as measured by the PROMIS psychological stress experience measure | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  PROMIS psychological stress experience measure is validated for pediatrics and adults. Scores range from 0-95 where 0 indicates no psychological stress and 95 is the maximum score for psychological stress.
Cognitive functioning, as measured by the PROMIS Cognitive Function Short Form for Adults and the PROMIS Cognitive Function Short Form for Pediatrics | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  PROMIS Cognitive Function Adult form scores range from 8-40, where 8 indicates never having cognitive dysfunction, and 40 indicates very often having cognitive dysfunction. PROMIS Cognitive Function Pediatric form scores range from 7-35, where 7 indicates never having cognitive dysfunction, and 35 indicates having cognitive dysfunction all of the time.
Quality of life, as measured by the Pediatric Quality of Life (PedsQL) Generic Core | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PedsQL measures quality of life in several aspects such as health, school, daily activities. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life.
Quality of life, as measured by the Pediatric Quality of Life (PedsQL) Rheumatology Core | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The PedsQL measures quality of life in several aspects such as pain and hurt, daily activities, treatment, worry, and communication. Each item is reversed scored and transformed to a linear scale of 0-100, such that 100 indicates a high quality of life and 0 indicates a low quality of life.
Medication adherence, as measured by the Medication Adherence Self-Report Inventory (MASRI) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The MASRI measures medication adherence on a scale of 0%-100%, such that lower scores indicate less adherence and higher scores indicate more adherence.
Disease activity, as measured by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The SLEDAI 2K measures disease activity in SLE, and takes into consideration descriptors of the disease such as arthritis and vasculitis. Higher scores indicate more active disease/flares, and lower scores indicated less disease activity.
Disease activity, as measured by the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The SLICC measures disease activity by assessing descriptors in SLE. Higher scores indicate greater disease activity, lower scores indicate lesser disease activity
Disease activity, as measured by the Lupus Low Disease Activity State (LLDAS) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The LLDAS is a score from 0-5, where 0 indicates higher disease activity state and 5 indicates lower disease activity state. The LLDAS includes 5 components, each receiving either a 1 (true) or a 0 (false): 1. SLEDAI score less than or equal to 4, 2. no new lupus disease activity, 3. a SELENA-SLEDAI less than or equal to 1, 4. a maintained low prednisolone dose, and 5. well tolerated maintenance doses or immunosuppressive drugs and approved biological agents.
Disease manifestations | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Disease manifestation will be assessed by use of the Systemic Lupus International Collaborating Clinics/ACR Damage Index for Systemic Lupus Erythematosus (SLICC) criteria checklist.
Anxiety, as measured by the Screen for Child Anxiety Related Disorders (SCARED) and Screen for Adult Anxiety Related Disorders (SCAARED) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The SCARED measures anxiety in children on a scale of 0 to 82, such that lower scores indicates low levels of anxiety, and high scores indicated high levels of anxiety. The SCAARED measures anxiety in adults on a scale of 0 to 88 such that lower scores indicated lower levels of anxiety and high scores indicate higher levels of anxiety. Both scales are comprised of sub-scales to measure types of anxiety (such as separation anxiety).

OTHER OUTCOMES:
Reach | April, 2023 to October, 2027
  Enrollment rates are the percent of patients enrolled. Reasons for not enrolling will also be collected.
Adoption | April, 2023 to October, 2027
  The number of champions using TEACH during active waves will be assessed.
Fidelity | April, 2023 to October, 2027
  Providers will be asked to create a registry of patients they see and those who are enrolled. They will be asked to keep data on how many patients complete each TEACH session (up to six). Format of session completion (in person vs. telehealth) and patient use of supplemental web support tools will also be explored.
Feasibility, acceptability, and appropriateness | April, 2023 to October, 2027
  Twelve psychometrically validated items to assess program feasibility, acceptability, and appropriateness, will be administered to champions after training. Patients and champions will rate items based on responses ranging from strongly agree (5) to strongly disagree (1) (scores ranging from 12-60, where 12 is low agreement and 60 is high agreement).
Provider knowledge | April, 2023 to October, 2027
  A pre/post a knowledge quiz self-reported items from a prior project evaluating knowledge of pediatric pain management strategies.
  Self-report items with five responses ranging from strongly agree (5) to strongly disagree (1) will also be used.
Implementation success | April, 2023 to October, 2027
  Qualitative interviews will be used to identify program feasibility, acceptability, appropriateness, and potential areas of refinement, barriers and facilitators of TEACH and measure implementation success with patients after TEACH is delivered.
Implementation success | April, 2023 to October, 2027
  Qualitative interviews will be used to identify program feasibility, acceptability, appropriateness, potential areas of refinement, barriers, and facilitators of TEACH and measure implementation success with mental health champions after they receive intervention training.
Maintenance | April, 2023 to October, 2027
  Monthly provider surveys to assess the number of patients who use TEACH clinically (after formal enrollment) will be collected during this phase. The number of patients (by site) who use the TEACH (number of sessions use, format, and use of web support tools) will also be collected. Data on whether champions train others in TEACH will also be collected.
Adverse Childhood Events (ACEs) | Through study completion, up to 56 weeks
  The ACEs questionnaire poses 9 different potential adverse childhood experiences in which participants indicate if they have or have not had that experience. The total is calculated by adding the items indicated as "yes."
Area Deprivation Index (ADI) | Baseline (T1)
  ADI will be used to assess neighborhood social disadvantage in United States participants, where >60% is defined as social deprivation.
Canadian Index of Multiple Deprivation (CIMD) | Baseline (T1)
  CMID will be used to assess neighborhood social disadvantage in Canadian participants, where >60% is defined as social deprivation.
Pubertal Development Scale | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Validated pubertal development scale will be given to participants regarding their physical development.
COVID-19 Diagnosis | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  To assess whether a patient has been or is currently diagnosed by COVID (and when).
Depression Anxiety and Stress Scales 21 (DASS21) (caregiver) | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  The DASS21 depression, anxiety, and stress on a scale of 0-63 with 0 indicating low levels of these feelings, and 63 indicating high levels. This measure will only be completed by caregivers participating in the study.
Concomitant medications | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Medications and vitamin/supplementation use will be collect through medical charts and reported by participants and caregivers of participants who are under 18 years.
Concomitant treatment | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Other treatments (therapies, massage, supplementation, etc.) will be reported by participants and caregivers of participants who are under 18 years.
Demographic information of participants | T1 (baseline), T2 (8 weeks), T3 (20 weeks), T4 (32 weeks), T5 (44 weeks), T6 (56 weeks)
  Patient age, sex, gender, race, ethnicity, family income, caregiver/patient education, zip code, and disease duration will be obtained.
Demographic information of mental health champions | T1 (baseline)
  Age, sex, gender, race, ethnicity, type of provider, years of practice, years on their current team, during of working with patients, site served
Adverse events | Throughout the duration of the study.
  Data on adverse events (study-related and non-study related) will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Natoshia R Cunningham, PhD, Principal Investigator — Michigan State University; Andrea Knight, MD, MSCE, Principal Investigator — The Hospital for Sick Children
Locations (7):
- United States (6):
  - University of Alabama Birmingham Hospital, Birmingham, Alabama
  - Children's Hospital of New Orleans/ Tulane University, New Orleans, Louisiana
  - Helen Devos Children's Hospital, Grand Rapids, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada